CLINICAL TRIAL: NCT05852405
Title: Clinical Characteristics, Natural History, Health Care Measures, and the Frequency of Genetic Variants in the Genes of SOD1, C9orf72, FUS and TARDBP in Patients With Sporadic and Familial Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Clinical Characteristics, Natural History, Health Care Measures, and Genetic Screening in Patients With ALS
Acronym: ID-ALS
Status: Completed | Type: Observational
Sponsor: Ambulanzpartner Soziotechnologie APST GmbH (Industry)
Collaborators: Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor
Other Study IDs: 400634
Record Dates: First submitted 2023-04-28; First posted 2023-05-10 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Motor Neuron Disease, Amyotrophic Lateral Sclerosis
Keywords: ID-ALS; ALSFRS-R-SE; ALSFRS-R; Neurofilament light chain NfL; APST Research; ALS-App; SOD1; C9orf72; FUS; TARDBP; Biomarker
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Frontotemporal Dementia With Motor Neuron Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — whole blood and serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with sporadic ALS (sALS), which refers to those without a family history of ALS, are typically not subjected to genetic investigations as part of their standard care. Therefore, their mutation status is often unknown. Even patients with familial ALS (fALS), who have a known family history of ALS, are not regularly screened for genetic mutations. This project aims to study a large group of ALS patients, examining their family history, clinical characteristics, healthcare measures, and genetic variants in ALS's most commonly mutated genes: SOD1, C9orf72, FUS, and TARDBP. Examining genetically distinct ALS cohorts is significant, as understanding the relationship between genotype and disease progression is essential in determining the therapeutic potential of future genetic therapies.

DETAILED DESCRIPTION:
Only limited data are available on the frequency of genetic variants in patients with sporadic ALS (sALS) and familial ALS (fALS). Genetic investigations do not belong to the standard of care in patients with sALS (patients without a family history of ALS). As a result, the patient's mutation status is commonly unknown. Even in patients with fALS (with a known family history of ALS), screening for genetic mutations is not performed regularly due to lacking treatment options in gene therapy. However, this paradigm is about to change as clinical trials on genetic medicines are ongoing and might result in the approval of new genetically investigated drugs. This project aims to explore a large cohort of ALS patients on family history, clinical characteristics, healthcare measures, and genetic variants in SOD1, C9orf72, FUS, and TARDBP - the most commonly mutated genes in ALS. This cohort study will allow us to determine the frequency of gene mutations in ALS patients in a real-world setting of ALS centers in Germany. Furthermore, the project shall enhance insights into potential differences between genetically defined cohorts using the course of the disease and the provision of health care measures. The investigation of genetically distinct ALS cohorts is particularly relevant, as an improved understanding of the relationship between the genotype and the journey of disease is scientifically indispensable to determine the therapeutic potential of future genetic therapies.

ELIGIBILITY:
Inclusion Criteria:

* ALS, including classical ALS, Progressive Muscle atrophy (PMA) or Primary Lateral Sclerosis (PLS)
* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) under national and local subject privacy regulations
* Age of 18 years old at the time of informed consent

Exclusion Criteria:

* Inability to provide patient directives about the notification of individual study results on genetic variants of SOD1, C9orf72, FUS and TARDBP
* Inability to comply with study requirements
* Unspecified reasons that, in the opinion of the site investigator, perceive the subject as unsuitable for enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The enrollment of subjects takes place in specialized ALS outpatient centers in Germany. ALS patients eligible for the investigation will be invited to participate in this cohort study. After obtaining informed consent, subjects will be enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Genetic variants in the genes of SOD1, C9orf72, FUS and TARDBP | 2 years
  • To identify the frequency of genetic variants in the genes of SOD1, C9orf72, FUS and TARDBP in patients with sALS and fALS

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Meyer, Prof. Dr., Study Director — Center for ALS and other motor neuron disorders, Charité - Universitätsmedizin Berlin
Locations (1):
- Center for ALS and other motor neuron disorders, Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-02): https://cdn.clinicaltrials.gov/large-docs/05/NCT05852405/Prot_SAP_000.pdf